CLINICAL TRIAL: NCT04955145
Title: Evaluation of The Effect of Rutin and Vitamin C on the Oxidative Stress in Hemodialysis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, samia mohamed omar, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUC-Fb-ASU RHDIRB2020110301
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: End Stage Renal Disease
Keywords: Oxidative stress, antioxidants, hemodialysis, vitamin C and Rutin
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ruta C 60 group (Active Comparator): Ascorbic Acid/Rutoside 60 tablet , each tablet contains: Rutin 60mg and Ascorbic acid 160mg Dosage:2 tablets three times daily for 4 months
  Interventions: Drug: RUTA C 60
- C- Retard group (Active Comparator): Ascorbic acid 500mg capsule dosage: 1 capsule two times daily for 4 months
  Interventions: Drug: RUTA C 60
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: RUTA C 60 — Rutin known as vitamin p or rotoside and C-retard is Ascorbic acid
  Other Names: C-retard
  Arms: C- Retard group; Ruta C 60 group

SUMMARY:
The aim of the study is to evaluate the effect of rutin and vitamin C on selected oxidative stress and inflammatory markrers.

Patients will be recruited according to the inclusion and exclusion criteria and will be divided into 3 groups, Group 1: Patients will administer a combination of Vitamin C and Rutin (RUTA C 60 tablets) in a dose of 2 tablets 3 times daily for 4 months in addition to their standard therapy, Group 2: will administer vitamin C 500mg hard gelatin capsules (twice daily) in addition to their standard therapy for a period of 4 months, Group3 (Control group) will administer the standard therapy. Blood samples will be withdrawn for measurement of; MDA, TNF-α ,GSH-PX, C-RP levels and ESR.

DETAILED DESCRIPTION:
Evaluation of the Effect of Rutin and Vitamin C on the Oxidative Stress in Hemodialysis Patients

A Protocol Submitted for Partial Fulfillment of Master Degree in Pharmaceutical Sciences (Clinical pharmacy)

By:

Samia mohamed omar

Under supervision of

Prof. Dr. Nagwa Ali Sabri Professor and head of clinical pharmacy department Faculty of pharmacy Ain shams university

Assoc. Prof. Tamer Wahid El Said Associate professor of Nephrology Faculty of medicine Ain shams university

Dr. Radwa Maher Abd-el-Kader-el-Borolossy Lecturer of Clinical Pharmacy Faculty of pharmacy Ain Shams University

Introduction

Morbidity and mortality are the most current important problems encountering medical scientists in the world in chronic kidney disease patients. (Kazi et al, 2008) Oxidative stress is associated with oxidative damage to proteins, lipids, and DNA and is playing an important role in disease progression in chronic kidney disease patients, in oxidative stress, reactive oxygen species(ROS) production exceeds the antioxidant capacity, also in hemodialysis, oxidative stress increased due to low-compatibility dialysis membrane treatments, which activates neutrophils and monocytes (phagocytic cells), and also due to a decrease in antioxidant capacity in which the activity superoxide dismutase, glutathione peroxidase, and peroxiredoxin2 enzymes is reduced in addition to low levels of non enzymatic antioxidants like vitamins C, E, and, A.(Gwozdzinski K et al, 2021) Several comorbidities in ESRD patients are related to oxidative stress characterized by high levels of pro-oxidants, like dyslipidemia, vascular calcification, hypertension, diabetes mellitus(DM), and old age.(Mondaresi et al, 2015) Malnutrition status, and chronic inflammation accompanies dialysis also triggers reactive oxygen species production.(handelman et al, 2001) 14 times increase in ROS levels is induced after each hemodialysis session.(Nguyen et al, 1985; Chen et al, 1998; Yang et al, 2006)

The kidney synthesizes the antioxidant enzymes , including glutathione peroxidases and its failure leads to reduced levels of these enzymes and as a consequence pro-oxidants are increased .(Kelly, Rothwell, 2020) The oxidation of fatty acids by free radicals is called lipid peroxidation and it is responsible for tissue damage.(Fatani et al, 2016) Malondialdehyde generated from lipid peroxidation is a nucleophilic agent has the ability to attack and change functions of amino acids and sulfhydryl moiety of proteins.(Slatter et al, 2000) Several studies have approved that enhanced rate of mortality in hemodialysis patients was associated with oxidative stress in relation with increased levels of MDA ,end product of unsaturated fatty acid oxidation.(Juretic et al, 2001) Antioxidants are endogenous antioxidants produced by the body (enzymatic and non enzymatic) and exogenous antioxidants present in food and supplements.(Liakopoulos et al, 2019) Vitamins B, C, D, and E,coenzymeQ10, L-carnitine, a-lipoic acid , curcumin, green tea, flavonoids, polyphenols, omega-3polyunsaturated fatty acid, statins, trace elements, and N-acetyl cysteine have been studied as exogenous antioxidants for reducing oxidative stress in hemodialysis patients.(Liakopoulos et al, 2019) Reducing oxidative stress in hemodialysis patients by using antioxidant treatments may be of useful approach in order to save life , to avoid death struggle, and to improve their quality of life19.(Navarro et al,2019) Many clinical studies present in databases have confirmed improved complications accompanied dialysis in patients supplemented with herbal antioxidants .(Asgharpour M, Alirezaei A , 2012) Lately, attention is increasing toward the antioxidant effect of rutin.( Moretti E et al, 2012)

Flavonoids has recently recognized by scientific group as a unique class of therapeutic molecules due to their various pharmacological properties, rutin, known as vitamin p or rotoside has been discovered for many of pharmacological effects.( Ganeshpurkar A, Saluja AK, 2017) Rutin is a flavonol , found in passion flower, buckwheat, tea, and apple.( Ganeshpurkar A, Saluja AK, 2017) Rutin called rotoside, quercetin-3-rutinoside, and sophorin is acitrus flavonoid glycoside.( Kreft S, Knapp M, Kreft I, 1999) Rutin is a phytochemical has many therapeutic properties . ( Ganeshpurkar A, Saluja AK, 2017) An ancient saying an apple a day, keeps doctor away appear to be right, as rutin, found in apples has many biological activities. ( Ganeshpurkar A, Saluja AK, 2017) Rutin is needed to be studied extensively to demonstrate effective safety profile in human to get its benefits as therapeutic supplement. ( Ganeshpurkar A, Saluja AK, 2017) Rutin as treatment was found to produce considerable impact on secretion of cytokines. ( Gandhi GR et al, 2020) Cytokines are secreted by immune cells, and inflammation during long term diseases, causes cytokines- mediated organ dysfunction and tissue damage, such as in diabetes mellitus, cancer, Rheumatoid arthritis. (Gautam R et al, 2006) The immunomodulatory and anti-inflammatory effects of rutin on chronic metabolic diseases support the idea that the rutin can be used in treating such these disorders and their complications. (Gandhi GR et al, 2020) Blood glucose reduced and lipid profile improved by using rutin, also activities of ALT, AST, and LDL in the liver, serum, and heart changes are prevented by rutin, rutin was found to has the ability to reduce hepatic and cardiac levels of TG and Enhances the glycogen level. (Gandhi GR et al, 2020)

Amazingly, the stability of rutin aganist oxidation was found to be greater than its aglycogen, quercetin. (Suzuki et al,2005) Rutin frequently used combined with vitamin C because it is essential for vitamin C absorption and as anti -oxidizer. (Bus ze Wski et al,1993) Human body cannot synthesize flavonoids and the diet can supply rutin, and rutin is not only for shelf-life prolongation of products, but also increases the nutritional value of products. (Chua LS, 2013) In addition to toxins hemodialysis removes nutrients from the blood, such as ascorbic acid (AA) and also hemodialysis patients are deficient from ascorbic acid due to dietary restrictions and this triggers oxidative stress and inflammation already induced by uremia ending with cardiovascular events and mortality.(Chaghouri P et al, 2021) ROS reduced by AA, particularly superoxide anion radical, and in turn ascorbic acid oxidized. (Bendich A et al, 1986) AA acid competitively reacts with ROS, scavenging them before they oxidize the cell components, and AA is oxidized, protecting lipid membranes, proteins, and DNA from damage. (Berratta M et al, 2020) In leukocytes ascorbic acid concentrations reaches 50-to100- higher than in plasma. (Berratta M et al, 2020) There are no studies conducted about the effect of rutin as antioxidant on the oxidative stress in hemodialysis patients.

Regarding the antioxidant and anti-inflammatory efficiency of AA, it is essential to see vitamin c effect on hemodialysis patients. (Chaghouri P et al, 2021) Relying on the antioxidant and anti-inflammatory effect of both, rutin and vitamin c confirmed by a variety of studies in vitro and in vivo rutin and vitamin C are selected to be studied in hemodialysis patients.

Aim of the study The aim of this study is to evaluate the effect of rutin and vitamin C on selected oxidative stress and inflammatory markers.

Patient and methods

1. Design:

   Prospective, interventional, Open label, randomized controlled clinical trial will be conducted on adult patients with ESRD on regular hemodialysis.
2. Settings:

The study will be carried out at nephrology and dialysis unit in ain shams university hospital

A total of 105 patients will be recruited and divided into 3 groups: - Group 1: (Ruta C group) 35 patients will take a dose of 2 tablets of rutin 60 mg in combination with vitamin C 160 mg three times daily for 4 months in addition to their standard therapy.

Group 2: (Vitamin C group) 35 patients will take a dose of 500mg of vitamin C two times daily for 4 months in addition to their standard therapy.

Group 3: Control group, 35patients will take only the standard therapy.

Baseline characteristics: The following data will be collected from all patients at baseline

1. Age, sex , weight, duration of ESRD and hemodialysis comorbidities .
2. Dialysis duration, BUN, Cr (mg/d L), Albumin (mg/d L), Hb (g m%), renal function test, liver function test, blood glucose level, TG, total cholesterol level, LDL-C, HLD-C.

Monitoring parameters:

1. Patients will be monitored for side effects.
2. blood sample will be withdrawn at baseline and at the end of the study from all groups then the sera will be centrifuged at 3000 rpm, for 10 minutes at 4°c, and then kept frozen at -80 C for the biochemical evaluation plasma malondialdehyde, C-Reactive Protein, GSH-PX, TNF-α and ESR. This analysis will be performed by enzyme linked immunosorbent assay technique (ELISA)

Ethics Consideration:

* The study will be performed according to Declaration of Helsinki.
* Approval of the Research Ethics committee of faculty of pharmacy - Ain-Shams university- faculty of pharmacy research ethics committee institutional review board.
* An Informed consent will be taken from all patients before enrollment in the study without any obligatory on the patients to withdraw from the study if they want to.

Statistical analysis:

Statistical analyses will be done using the SPSS software (Statistical Package for the Social Sciences). Continuous variables will be represented as mean + standard deviation (SD) or as median + interquartile range (IQR). Statistical tests will be chosen based on either the resulting data will be parametric or non-parametric. P-values lower than 0.05 are considered statistically significant and P-values lower than 0.001 are considered highly significant.

Sample size calculation:

The sample size was calculated by GPower v.3.1.9.4 1. According to Connelly (2008), the literature suggests that a pilot study sample should be 10% of the sample 3 equally sized groups and an alpha of 0.05, the sample size would be 966 participants. For our pilot study, the required sample size would be 97 participants. To account for dropouts and projected for the larger parent study 2.

Therefore, for a full-scale study, expecting a small effect size of 0.10, to reach a power of 80% to reject the null hypothesis, with equality of group sizes, we decided to recruit a total of 105 participants, equally divided among the 3 groups (35 participants in each group).

F tests - ANOVA: Fixed effects, omnibus, one-way Analysis: A priori: Compute required sample size Input: Effect size f = 0.10 α err prob = 0.05 Power (1-β err prob) = 0.80 Number of groups = 3 Output: Noncentrality parameter λ = 9.6900000 Critical F = 3.0050418 Numerator df = 2 Denominator df = 966 Total sample size = 969 Actual power = 0.8011010

ELIGIBILITY:
Inclusion Criteria:

* Age of patients > 18 year old.
* hemodialysis in the last 3 months or longer.
* hemodialysis frequency 3 times per week or more.

Exclusion Criteria:

1. Treatment with antioxidant agents [such as vitamin C and E during the 2 preceding months prior to the study.
2. Active liver disease
3. pregnant patients or patients planning pregnancy.

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
The change in Malondialdehyde(MDA) level from the baseline will be assessed at the end of the study (after the end of the intervention) | At baseline(pre-intervention)
  Micromole/L
The change of Malondialdehyde(MDA) level from the baseline(Pre-intervention) will be assessed at the end of the study (after the end of the intervention) | At end of the study (After the end of the intervention immediately)
  Micromole/L
The change of Glutathione peroxidase(GSH-PX) level from the baseline will be assessed at end of the study(After end of the intervention) | At baseline(pre-intervention)
  Micromole/L
The change of Glutathione peroxidase(GSH-PX) level from the baseline(pre-intervention) will be assessed at end of the study(After end of the intervention immediately) | At end of the study (After the end of the intervention immediately)
  Micromole/L
The change of Tumor necrosis factor-alpha(TNF-alpha) level from the baseline will be assessed at the end of the study (after the end of the intervention immediately) | At baseline(pre-intervention)
  pg/ml
The change of Tumor necrosis factor-alpha(TNF-alpha) level from the baseline will be assessed at the end of the study | At end of the study(After the end of the intervention immediately)
  pg/ml
The change of C-Reactive protein(C-RP) level from the baseline will be assessed at the end of the study | At baseline(pre-intervention)
  mg/L
The change of C-Reactive protein(C-RP) level from the baseline will be assessed at the end of the study | At end of the study(After the end of the intervention immediately)
  mg/L
The change in Erythrocyte sedimentation rate from the baseline will be assessed at the end of the study Erythrocyte sedimentation rate (ESR) | At baseline(pre-intervention)
  mm/hour
The change in Erythrocyte sedimentation rate from the baseline will be assessed at the end of the study | At end of the study(After the end of the intervention immediately)
  mm/hour

SECONDARY OUTCOMES:
Quality of life of end stage renal disease patients on hemodialysis | At baseline(pre-intervention)
  The Kidney Disease Quality of Life short form questionnaire 36 Physical function Physical role Pain General health Physical component summary Emotional well-being Emotional role Social function Energy/fatigue Mental component summary Symptoms and problems Effects of kidney disease Burden of kidney disease Work status Cognitive function Quality of social interaction Sexual function Sleep Social support Dialysis staff encouragement Patient satisfaction Kidney disease component summary
  SF, short form. For each domain and, summary measure, the score ranges from 0 to 100, with a higher score indicating better quality of life.
Quality of life of end stage renal disease patients on hemodialysis | At end of the study(After the end of the intervention immediately)
  The Kidney Disease Quality of Life short form questionnaire 36 Physical function Physical role Pain General health Physical component summary Emotional well-being Emotional role Social function Energy/fatigue Mental component summary Symptoms and problems Effects of kidney disease Burden of kidney disease Work status Cognitive function Quality of social interaction Sexual function Sleep Social support Dialysis staff encouragement Patient satisfaction Kidney disease component summary
  SF, short form. For each domain and, summary measure, the score ranges from 0 to 100, with a higher score indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Samia Mohamed Omar, Master student, Principal Investigator — Faculty of pharmacy-Ain shams university
Locations (1):
- Ain shams university hospitals, Cairo, Egypt